CLINICAL TRIAL: NCT01497223
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Study of Fluconazole Versus Fluconazole And MGCD290 for the Treatment of Moderate to Severe Vulvovaginal Candidiasis
Brief Title: MGCD290 and Fluconazole Versus Fluconazole Alone for the Treatment of Moderate to Severe Vulvovaginal Candidiasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MethylGene Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 290-005
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2012-06

CONDITIONS: Vulvovaginal Candidiasis
Keywords: Phase II; Double-Blind; Placebo-Controlled; Vulvovaginal Candidiasis; Moderate to Severe; Acute; Treatment of Moderate to Severe Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MGCD290 and Fluconazole (Experimental): Oral Administration of MGCD290 and Fluconazole
  Interventions: Drug: MGCD290
- Fluconazole (No Intervention): This is an Active Comparator: Oral Administration of Fluconazole with Placebo

INTERVENTIONS:
Drug: MGCD290 — 1 Oral Dose Administration
  Arms: MGCD290 and Fluconazole

SUMMARY:
The primary objective of the study is to evaluate the rate of therapeutic cure of the combination treatment of MGCD290 and fluconazole as compared to that of fluconazole alone at Test of Cure Visit for patients with moderate to severe vulvovaginal candidiasis.

DETAILED DESCRIPTION:
MGCD290 is a novel antifungal agent targeting the Hos2 enzyme in fungi. MGCD290 was shown to potentiate and broaden the spectrum of activity of azole antifungal agents in vitro, especially fluconazole. MGCD290 taken together with fluconazole was observed to be safe in healthy volunteer studies. The current study is evaluating both the efficacy and safety of the combination treatment in subjects with moderate to severe vulvovaginal candidiasis.

ELIGIBILITY:
Inclusion Criteria:

* Vulvovaginal candidiasis infection is diagnosed, the symptoms evaluated using a numerical rating system based on severity (absent=0; mild=1; moderate=2; severe=3) with a minimum VVC Composite Signs/Symptoms score of 7.
* Subject with normal vaginal pH (≤4.5) upon evaluation.
* Subject completes the informed consent process.
* Subject agrees to take study medication when scheduled. Subject has no difficulty swallowing the medication.
* Subject complies with all clinical trial instructions. Commits to all follow-up visits.
* Subject is free of any disease or physical condition which might impair the evaluation of safety and/or vulvovaginal candidiasis.
* Subject of childbearing potential has a negative urine pregnancy test at screening.
* Subject of childbearing potential agrees to use an effective, non-prohibited form of birth control for the duration of clinical trial or until onset of menses following the administration of study medication, whichever is longer. She must be on a stable regimen of oral contraceptives, contraceptive implant or depot injection, contraceptive patch, IUD, condom and spermicidal agent, diaphragm and spermicidal agent, or sexual abstinence for at least the past 60 days.
* Subject agrees to abstain from sexual intercourse from the time of randomization through the first seven days immediately following treatment.
* Direct microscopic examination with KOH must be positive at screening showing yeast forms (hyphae/pseudohyphae) or budding yeasts.
* Aged 18 and over, post-menarcheal, and not surgically or naturally post-menopausal.

Exclusion Criteria:

* Sensitivity to ingredients in the study medications.
* Subject currently participates in, or has within 30 days prior to this clinical trial participated in, an investigational clinical trial.
* Subject experienced 4 or more episodes of VVC in the past 12 months.
* Subjects with other causes of vulvovaginitis.
* Subjects with active HPV infection.
* Subjects with other urogenital infections that would potentially alter their response to disease.
* Subjects with confirmed Neisseria gonorrhea or Chlamydia trachomatis.
* Subjects with abnormal PAP test results except for ASC-US with confirmed absence of High-Risk HPV infection.
* Subjects who will be under treatment or have surgery during the study period for cervical intraepithelial neoplasia or cervical carcinoma.
* Subjects with a planned major surgery during the time of the study.
* Pregnant or nursing subjects.
* Subjects menstruating at enrollment.
* History of hypersensitivity to azoles.
* Evidence/history of ventricular dysfunction such as congestive heart failure, unstable coronary artery disease, significant cardiac arrhythmias or proarrhythmic conditions associated with prolongation of QT interval.
* History of clinically significant ECG abnormalities, including QTc prolongation.
* Current treatment with: erythromycin, astemizole, pimozide, quinidine, and cisapride)
* History of cancer or currently being treated for a cancer.
* Subject is immunocompromised or has chronic mucocutaneous candidiasis.
* Use of systemic immunosuppressants such as cyclosporine, TNF inhibitors and tacrolimus.
* History of liver toxicity with other drugs.
* History of hepatic or renal impairment.
* Subjects with diabetes mellitus with poor glycemic control (HgbA1C >7%).
* Subjects with any other concurrent significant uncontrolled illness.
* Use of oral antifungals within 14 days immediately prior to enrollment.
* Use of systemic corticosteroids within 30 days immediately prior to enrollment (inhaled corticosteroids are permitted).
* Use of any topical vaginal products within 1 week prior to enrollment.
* Subject is a substance abuser such that the abuse may result in lack of study compliance.
* Vaginal pessaries and rings used for contraception or hormone replacement therapy.
* Subject used an antibiotic within 24 hours immediately prior to enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Therapeutic Cure Rate | 28 Days

SECONDARY OUTCOMES:
Mycological Cure Rate | Day 14 and Day 28
Clinical Cure Rate | Day 14 and Day 28
Therapeutic Cure Rate | Day 14
Recurrence Rate | Day 28
Time to Resolution of Symptoms | First 14 days post-dose
Improvement in Symptoms | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reid, MSc, MBA, Study Director — MethylGene Inc.
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Women's Health Care Research Corp., San Diego, California
  - Altus Research, Lake Worth, Florida
  - Healthcare Clinical Data, Inc., North Miami, Florida
  - Georgia Health Sciences University, Augusta, Georgia
  - Clinical Trials Management, Covington, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Harper University Hospital, Detroit, Michigan
  - Clinical Research of Nevada, Las Vegas, Nevada
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Lyndhurst Clinical Research, Raleigh, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Brownstone Clinical Trials, Irving, Texas
  - Physician's Research Options, Sandy City, Utah
  - Tidewater Physicians for Women, Norfolk, Virginia
  - University of Washington, Seattle, Washington